CLINICAL TRIAL: NCT02020395
Title: Effect of a Test Meal on Satiation Hormones in Obese and Normal Weight Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GI peptides obese adolescents
Record Dates: First submitted 2013-12-12; First posted 2013-12-24 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Endocrine System Diseases
MeSH Terms: conditions — Endocrine System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test meal (500 kcal)_normal weight (Placebo Comparator): ham sandwich chocolate cream orange juice
  Interventions: Dietary Supplement: test meal (500 kcal)
- Test meal (500 kcal)_obese weight (Active Comparator): ham sandwich chocolate cream orange juice
  Interventions: Dietary Supplement: test meal (500 kcal)

INTERVENTIONS:
Dietary Supplement: test meal (500 kcal) — whole wheat bread (68 g), butter(10 g), ham (25 g); chocolate cream (90 g); orange juice (200 mL)
  Arms: Test meal (500 kcal)_normal weight
Dietary Supplement: test meal (500 kcal) — whole wheat bread (68 g), butter(10 g), ham (25 g); chocolate cream (90 g); orange juice (200 mL)
  Arms: Test meal (500 kcal)_obese weight

SUMMARY:
The objective of this study is to examine ghrelin, amylin, glucagon and glucagon-like peptide (GLP)-1 responses to a test meal in lean and obese individuals.

DETAILED DESCRIPTION:
The primary hypothesis is that obese adolescents have a disturbed balance of hormones associated with appetite regulation with less suppression of ghrelin and attenuated stimulation of GLP-1 secretion in response to meal intake compared to lean normal weight controls. A second aim of the study was to test which gastrointestinal peptides are most associated with insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* caucasian youth
* pubertal Tanner stage x, y, or z

Exclusion Criteria:

* fasting plasma glucose > 7.0 mmol/L
* significant illness
* taking medications

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Comparison of gastrointestinal peptide secretion in normal weight and obese adolescents | 2 hours blood sampling
  Relation of GLP-1 release to insulin secretion in normal weight and obese adolescents

SECONDARY OUTCOMES:
Association between gastrointestinal peptides and insulin release | 2 hours blood sampling
  Dynamics of gastrointestinal peptide secretion including Tmax and Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Principal Investigator — Division of Gastroenterology and Hepatology, University Hospital Basel
Locations (1):
- University Hospital Basel, Division of Gastroenterology and Hepatology, Basel, Switzerland